CLINICAL TRIAL: NCT06529289
Title: Effectiveness of Female Community Health Volunteers Training Program on Hypertension Knowledge and Blood Pressure Measurement Skills in Kavrepalanchowk, Nepal
Brief Title: Effectiveness of Female Community Health Volunteers Training on Hypertension Knowledge and Blood Pressure Measurement Skills in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Archana Shrestha, Associate Professor, Kathmandu University School of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 36/24
Record Dates: First submitted 2024-07-23; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Female Community Health Volunteers
Keywords: Effectiveness; Training; Hypertension; Knowledge; Blood Pressure Measurement Skills
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training to Female Community Health Volunteers (Other): Female Community Health Volunteers received a one-day training on hypertension knowledge and blood pressure measurement skills. The training included sessions on hypertension knowledge and practical demonstrations of BP measurement techniques. The effectiveness of the training was assessed by measuring the baseline and end-line hypertension knowledge and BP measurement skills."
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — We conducted one day of training for FCHVs and four different groups of FCHVs from two municipalities. We conducted training on hypertension knowledge and blood pressure measurement skills for FCHVs. Studies from Nepal show that with appropriate training, FCHV has the potential to promote hypertension education and conduct hypertension screening. Access to essential equipment such as digital blood pressure monitors, would improve FCHV performance on measuring blood pressure. Therefore, our training was to provide hypertension knowledge and to train FCHVs to measure blood pressure.
  The training had two objectives referring to enhancing knowledge and building skills.

SUMMARY:
The investigators aimed to investigate the effectiveness of training FCHVs in hypertension knowledge and blood pressure measuring skills and explore their perceptions of challenges and opportunities to deliver hypertension counseling and monitor Blood pressure in the community. The investigators conducted a quasi-experimental study design among 131 FCHVs from Namobuddha and Mandandeupur municipalities. The investigators quantitatively measured the baseline and end-line hypertension knowledge and BP measurement skills after providing a one-day training on hypertension knowledge and BP measurement. Furthermore, the investigators conducted three focus group discussions with FCHVs to explore the challenges and opportunities of FCHVs in community-based hypertension management.

DETAILED DESCRIPTION:
Female Community Health Volunteers (FCHVs) in Nepal could play a role in preventing and managing hypertension. Limited studies have been conducted on Nepal's FCHV knowledge and capacity to deliver hypertension-related counseling and services. The investigators investigate the effectiveness of training FCHVs in hypertension knowledge and blood pressure measuring skills and explore their perceptions of challenges and opportunities to deliver hypertension counseling and monitor Blood pressure in the community. The investigators conducted a quasi-experimental study design among 131 FCHVs from Namobuddha and Mandandeupur municipalities. The investigators quantitatively measured the baseline and end-line hypertension knowledge and BP measurement skills after providing a one-day training on hypertension knowledge and BP measurement. The investigators used the Hypertension Knowledge Level Scale (HK-LS) to assess the knowledge through face-to-face interviews and observed BP measurement skills using an observation checklist. The investigators used paired t-tests to see the mean difference before and after the training. The investigators performed linear regression to assess the hypertension knowledge and BP measurement skills scores with socio-demographic and FCHV's general performance. Furthermore, the investigators conducted three focus group discussions with FCHVs to explore the challenges and opportunities of FCHVs in community-based hypertension management. The investigators transcribed the recorded discussion verbatim and analyzed it using the framework analysis method

ELIGIBILITY:
Inclusion Criteria:

* Appointed as FCHV
* Age 18 years and older

Exclusion Criteria:

* Not able to respond during the data collection period
* Out of municipality during the data collection period

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Hypertension Knowledge | Baseline and endline data collected within a single day. 1 day
  We measured the FCHVs Hypertension in terms of knowledge score The Hypertension Knowledge Level Scale (HK-LS) assessed respondents' knowledge in defining hypertension, lifestyle, medical treatment, drug compliance, diet, and complications of hypertension. Each item was a complete sentence that was either correct or incorrect. Each item was prepared as part of a standard answer (correct, incorrect, or do not know). The scale included 22 items divided into six subdimensions (annex - IV). Each correct answer is worth 1 point. The maximum score is 22 for the entire scale. The minimum score is zero for the whole scale, and a score of higher means better knowledge for all sub-dimensions.

SECONDARY OUTCOMES:
Blood Pressure measurement skills | Baseline and endline data collected within a single day. 1 day
  Blood pressure skills were observed in three pre- and post-observation segments using an observational checklist. At first, pre-observation was performed, and training to measure blood pressure was provided to FCHVs; after that, post-observation was performed. There were pre-measurement inquiries and instructions for five items, measurement instructions for items, and a post-measurement record of 1 item. We ticked "yes" or "no" if the FCHV performed the activity listed in the checklist. Each 'yes' item gets 1 point, and the total score ranges from 0 to 17, with higher scores indicating a higher skill level. We defined blood pressure measurement capacity as an indicator of the FCHVs could perform these four actions: Placement of measuring arm at the level of heart, Proper fastening of the cuff, Measuring blood pressure three times at 1 (or more) minute(s) intervals, Recording of all readings).

CONTACTS AND LOCATIONS:
Overall Officials: Archana Shrestha, Principal Investigator — Kathmandu University School of Medical Sciences
Locations (1):
- Prasansha Poudel, Dhulikhel, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tan J, Xu H, Fan Q, Neely O, Doma R, Gundi R, Shrestha B, Shrestha A, Shrestha S, Karmacharya B, Gu W, Ostbye T, Yan LL. Hypertension Care Coordination and Feasibility of Involving Female Community Health Volunteers in Hypertension Management in Kavre District, Nepal: A Qualitative Study. Glob Heart. 2020 Oct 23;15(1):73. doi: 10.5334/gh.872. PMID 33150138
- [Result] Erkoc SB, Isikli B, Metintas S, Kalyoncu C. Hypertension Knowledge-Level Scale (HK-LS): a study on development, validity and reliability. Int J Environ Res Public Health. 2012 Mar;9(3):1018-29. doi: 10.3390/ijerph9031018. Epub 2012 Mar 22. PMID 22690180